CLINICAL TRIAL: NCT00359697
Title: Prospective, Randomized Clinical Trialto Compare Mannitol and Hypertonic Saline for Treatment of Increased Intracranial Pressure
Brief Title: Comparison of Two Different Medications Used to Treat Elevated Intracranial Pressure
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06U.132
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Increased Intracranial Pressure
MeSH Terms: conditions — Intracranial Hypertension | interventions — Saline Solution, Hypertonic; Mannitol

INTERVENTIONS:
Drug: Hypertonic Saline, Mannitol

SUMMARY:
The overall purpose of this study is to compare the effects of mannitol and hypertonic saline on patients with increased intracranial pressure. The hypothesis being tested is that hypertonic saline is more effective in controlling increased intracranial pressure than mannitol.

ELIGIBILITY:
Inclusion Criteria:

* Documented SAH (by computed tomography or lumbar puncture), ICH, TBI or brain tumor
* Patient greater than or equal to 18 years of age
* ICP monitor in place
* ICP greater than 20mmHg, not related to a transient noxious stimulus and not responding to standard measures for controlling ICP (ventricular drainage, elevation of head of the bed and optimizing PaCO2)
* Patient or patient's legally authorized representative has provided written informed consent

Exclusion Criteria:

* Patient less than 18 years of age
* Lack of ICP monitoring
* Patient received Mannitol prior to placement of ICP monitor
* Baseline serum osmolarity of greater than 310 mOsm/L
* Patient is currently enrolled in another investigational drug or device study
* Congestive heart failure at time of enrollment
* Chronic renal failure on hemodialysis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)

PRIMARY OUTCOMES:
Reduction of ICP below treatment threshold (less than 20 mmHg)

SECONDARY OUTCOMES:
Compare effects of each treatment on MAP, CPP, serum and urine sodium and osmolality

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Rosenwasser, MD, Principal Investigator — Thomas Jefferson University